CLINICAL TRIAL: NCT02222441
Title: A Phase 1, Open-label, Fixed-sequence, 2-cohort, 2-period Study To Investigate The Effect Of Modafinil And Pioglitazone Given As Multiple Doses On Single Dose Pharmacokinetics Of Palbociclib (Pd-0332991) In Healthy Volunteers
Brief Title: Effect Of Modafinil And Pioglitazone On The Pharmacokinetics Of Palbociclib (PD-0332991)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481039
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Palbociclib; Modafinil; Pioglitazone; Pharmacokinetics; Drug-Drug Interaction Study; Healthy Volunteers; CYP3A Inducers
MeSH Terms: interventions — palbociclib; Modafinil; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed sequence modafinil DDI arm (Cohort 1) (Experimental): Fixed sequence study with treatment A of palbociclib alone, followed by treatment B of palbociclib with modafinil in Cohort 1.
  Interventions: Drug: Palbociclib alone; Drug: Palbociclib plus Modafinil
- Fixed sequence pioglitazone DDI arm (Cohort 2) (Experimental): For Cohort 2, fixed sequence study with treatment A of palbociclib alone, followed by treatment C of palbociclib with pioglitazone.
  Interventions: Drug: Palbociclib alone; Drug: Palbociclib plus pioglitazone

INTERVENTIONS:
Drug: Palbociclib alone — A single 125 mg dose of palbociclib free base capsule given orally alone in the fed state, followed by 120 hours of PK sample collection.
  Other Names: Palbociclib, PD-0332991
  Arms: Fixed sequence modafinil DDI arm (Cohort 1)
Drug: Palbociclib plus Modafinil — For Cohort 1, modafinil 200 mg once daily for 7 days, followed by 400 mg once daily for 25 days; on Day 28, a single oral 125 mg dose of palbociclib will be given with modafinil after a meal, followed by 120 hours of PK sample collection.
  Other Names: Palbociclib (PD-0332991); Modafinil (Provigil)
  Arms: Fixed sequence modafinil DDI arm (Cohort 1)
Drug: Palbociclib alone — A single 125 mg dose of palbociclib free base capsule given orally alone in the fed state, followed by 120 hours of PK sample collection.
  Other Names: Palbociclib, PD-0332991
  Arms: Fixed sequence pioglitazone DDI arm (Cohort 2)
Drug: Palbociclib plus pioglitazone — For Cohort 2, pioglitazone 45 mg once daily for a total of 19 days; On Day 15, a single oral 125 mg dose of palbociclib will be given with pioglitazone after a meal, followed by 120 hours of PK sample collection.
  Other Names: Palbociclib (PD-0332991); Pioglitazone (Actos)
  Arms: Fixed sequence pioglitazone DDI arm (Cohort 2)

SUMMARY:
This study is designed to evaluate the potential effect of the moderate CYP3A inducer modafinil and the weak CYP3A inducer pioglitazone on the pharmacokinetics of palbociclib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Subjects with a self-reported history of addiction, especially to stimulants.
* A positive urine drug screen or alcohol breath test.
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-120 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0-120 hours

SECONDARY OUTCOMES:
Plasma Palbociclib Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 120 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Plasma Palbociclib Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0 to 120 hours
Plasma Palbociclib Decay Half-Life (t1/2) | 0 to 120 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) of Palbociclib | 0 to 120 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) of Palbociclib | 0 to 120 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Trough Plasma Concentrations of Modafinil, Modafinil sulfone, pioglitazone, hydroxy derivative of pioglitazone, and keto derivative of pioglitazone | 0 to 120 hours
Time of last quantifiable concentration for palbociclib | 0 to 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481039&StudyName=Effect%20Of%20Modafinil%20And%20Pioglitazone%20On%20The%20Pharmacokinetics%20Of%20Palbociclib%20%28PD-0332991%29